CLINICAL TRIAL: NCT03235505
Title: Efficacy and Safety of E-cigarettes for Smoking Cessation in Middle-aged Heavy Smokers
Acronym: EFFECT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oulu (Other)
Collaborators: Lapland Central Hospital Rovaniemi Finland (Unknown)
Responsible Party: Principal Investigator, Tuula Toljamo, MD, PhD, Chief Chest Physician of Lapland Central Hospital, University of Oulu
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WI218780
Record Dates: First submitted 2017-06-02; First posted 2017-08-01 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Smoking Cessation; Electronic Cigarette
Keywords: Smoking Cessation; Electronic cigarette; Adults
MeSH Terms: conditions — Smoking Cessation; Vaping | interventions — Nicotine; Varenicline; Motivational Interviewing

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Nicotine containing e-cigarettes (Experimental): Nicotine containing e-cigarettes + placebo-varenicline + Motivational Interview (MI)
  Interventions: Drug: Nicotine
- Nicotine-free e-cigarettes (Active Comparator): Nicotine-free e-cigarettes + varenicline tartrate+ MI
  Interventions: Drug: Varenicline Tartrate
- Motivational Interview (MI) (Placebo Comparator): Placebo-varenicline + nicotine -free e-cigarettes + MI
  Interventions: Behavioral: Motivational Interview

INTERVENTIONS:
Drug: Nicotine — Nicotine containing e-cigarettes + placebo-varenicline + Motivational Interview (MI)
  Other Names: Innokin Endura T20S
  Arms: Nicotine containing e-cigarettes
Drug: Varenicline Tartrate — Varenicline + Innokin Endura T20S electronic inhaler but without any nicotine content + MI
  Other Names: Champix
  Arms: Nicotine-free e-cigarettes
Behavioral: Motivational Interview — Placebo-varenicline + Innokin ENdura T20S electronic inhaler but without any nicotine content +MI
  Arms: Motivational Interview (MI)

SUMMARY:
Abstract Rationale. Electronic cigarette use is increasing at an exponential rate in Finland and internationally. The health consequences of vaporised aerosols in electronic cigarettes are largely unknown especially in a long run. Still, very few studies are available on quitting attempts with e-cigarettes as a smoking cessation tool compared to evidence based cessation pharmacotherapy in adult smokers who want to quit.

Research Objective: To investigate effectiveness and safety of e-cigarettes for smoking cessation in middle-aged smokers, and to compare the effectiveness of them to varenicline. Our study provides new information of success in smoking cessation among heavy adult smokers for clinicians.

Design: A double-blind, randomised, placebo-controlled clinical trial with the intervention phase of 12 weeks and the observational phase up to 52 weeks. This is an investigator initiated study.

Setting: Volunteer middle-aged daily smokers, who were recruited through newspaper announcements. Some of the cohort subjects were re-recruited from our previous follow-up study as many of them continued daily smoking during the whole follow-up period.

Participants: Targeted sample size of 450 adult heavy smokers, who want to quit smoking and are willing to participate up to 52 weeks´ follow-up.

Intervention and procedures: Standardized self-reported questionnaires with detailed smoking history with assessment of motivation to quit smoking, parameters of nicotine dependence, symptoms will be included. Smoking status will be repeatedly reassessed during the study visits, and self-reported smoking abstinence is verified with exhaled-carbon monoxide (CO) assessment. All adverse side effects either of drugs or of e-cigarettes, and symptoms related to the drugs or to withdrawal from smoking will be carefully reported.

DETAILED DESCRIPTION:
This is a study with three arms. Each arm has 12 weeks intervention and observation up to 12 months:

A.Nicotine containing e-cigarettes + placebo-pills + Motivational Interview (MI)

Innokin Endura T20S + USB cable with wall adapter via USB cable (output DC5V)+ + 6x 10ml /month refill containing 18mg/ml nicotine with cigarette taste for 12 weeks.

Participants are allowed to use ad libitum e-cigarettes during 12 weeks after they have chosen the quit day during the 2nd follow-up week

Placebo -pills: starting week: 0,5mg once daily on days 1.-3 and 0,5mg twice daily on days 4.-5.Continuing weeks: 1mg twice daily up to 12 weeks

B.Nicotine-free e-cigarettes + varenicline + MI

Innokin Endura T20S + USB cable with wall adapter via USB cable (output DC5V)+ + 6x 10ml /month refill containing 0mg/ml nicotine with cigarette taste for 12 weeks Participants are allowed to use ad libitum e-cigarettes during 12 weeks after they have chosen the quit day during the 2nd follow-up week

Varenicline (Chantix®) Starting week: 0,5mg once daily on days 1.-3 and 0,5mg twice daily on days 4.-5. Continuing weeks: 1mg twice daily up to 12 weeks

C.Placebo-varenicline + nicotine -free e-cigarettes + MI Placebo -pills : starting week: 0,5mg once daily on days 1.-3 and 0,5mg twice daily on days 4.-5.Continuing weeks: 1mg twice daily up to 12 weeks

Innokin Endura T20S + USB cable with wall adapter via USB cable (output DC5V)+ 6x 10ml /month refill containing 0mg/ml nicotine with cigarette taste for 12 weeks Participants are allowed to use ad libitum e-cigarettes during 12 weeks after they have chosen the quit day during the 2nd follow-up week

ELIGIBILITY:
Inclusion Criteria:

* Aged between 25 to under 75 years
* Has smoked over 10 years on a daily basis and being a current smoker with at least 10 cig/day for at least past 5 years
* Good general health
* Intent to quit smoking
* Exhaled carbon monoxide level at least 15ppm at the baseline visit
* Strong nicotine dependence defined by Fagerström Test for Nicotine Dependence (FTND) ≥ 5 and by Heaviness of Smoking Index (HSI) ≥3
* intent to quit smoking
* prepared to follow the trial protocol and able to provide written consent.

Exclusion Criteria:

* Pregnancy or gestation or intend to get pregnant during the study follow-up
* Use of smoking cessation pharmacotherapy or ECs during the past year
* Attempt of smoking cessation by using of e-cigarettes during the past year
* Any cancer (at least five healthy follow-up years after stopping the cancer therapy)
* Instable (ischemic) vascular or heart disease
* Recent myocardial infarction in the past three months
* High blood pressure (systolic BP> 140mmHg or diastolic 90mmHg at rest)
* History of major psychiatric depression or other psychiatric conditions and daily use of any psychiatric medicine
* Current addiction of alcohol or misuse of substance
* Inability to express himself/herself
* Known allergy to any of the study medications
* Severe allergy or poorly controlled asthma or other pulmonary disease
* Epilepsy

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Smoking cessation during the follow-up visit at week 26 | 24 week
  7-day point prevalence verified by exhaled-CO<10ppm

SECONDARY OUTCOMES:
Smoking cessation at any other study visit | Baseline,1, 12 and 52 week
  7-day point prevalence verified by exhaled-CO < 10pp
Reduce smoking at any study visit | Baseline, 1,4 ,12,16, 26, 36 and 52 week
  Prevalence of those who succeeded to decrease the number of daily cigarettes during the study

CONTACTS AND LOCATIONS:
Overall Officials: Tuula Toljamo, PhD, Principal Investigator — Laplnd Central Hospital Rovaniemi Finland
Locations (1):
- Lapland Central Hospital, Rovaniemi, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tuisku A, Rahkola M, Nieminen P, Toljamo T. Electronic Cigarettes vs Varenicline for Smoking Cessation in Adults: A Randomized Clinical Trial. JAMA Intern Med. 2024 Aug 1;184(8):915-921. doi: 10.1001/jamainternmed.2024.1822. PMID 38884987